CLINICAL TRIAL: NCT00407420
Title: Can a Novel Treatment Using "Mandometer®" Technology Improve Weight Loss in a Childhood Obesity Clinic?
Brief Title: "Mandometer®" Study for Managing Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bristol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJ4316
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Results first posted 2019-09-30 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Childhood Obesity
Keywords: Childhood; Obesity; Behavior modification; Insulin resistance
MeSH Terms: conditions — Pediatric Obesity; Obesity; Insulin Resistance

ARMS (2):
- Mandometer (Experimental): Active intervention - one meal eaten per day off Mandometer
  Interventions: Device: Mandometer; Behavioral: Lifestyle
- Control (Active Comparator): Nutritional and activity advice alone
  Interventions: Device: Mandometer

INTERVENTIONS:
Device: Mandometer — A computerised device, Mandometer, providing real time feedback to participants during meals to slow down speed of eating and reduce total intake; standard lifestyle modification therapy.
Behavioral: Lifestyle — Typical dietary and activity advice as normally provided in clinic (control).
  Arms: Mandometer

SUMMARY:
We run a successful clinic in Bristol for children with severe obesity who already demonstrate many features to suggest they are at increased risk of early diabetes and heart disease. However, we have found that young children respond better to simple interventions than do adolescents. We have used a new treatment regimen "Mandometer®" to help our most difficult adolescent cases lose weight. We would like to do a study to see if all adolescents might improve weight loss using this technology compared to what we routinely offer

DETAILED DESCRIPTION:
Childhood obesity is rapidly reaching epidemic proportions in the United Kingdom. Recent studies have indicated a prevalence level for obesity of 15% at 15 years of age. The implications for metabolic, cardiovascular and cancer risk in later life are enormous. The International Obesity Task Force (IOTF) and the European Association for the Study of Obesity (EASO) have identified childhood obesity as a matter for urgent attention. However, there are very few obesity clinics for children in the UK and effective treatment regimens are simply not available. We have developed an obesity clinic at the Royal Hospital for Children in Bristol and observed effective weight reduction in pre-pubertal children. Our simple treatment framework has proved far less effective in adolescence. We have therefore collaborated with an eating disorder clinic from the Karolinska Institute in Sweden to develop a novel therapy to treat obesity using modified equipment originally designed to treat adolescents with DSM-IV eating disorders. Pilot data indicate that adolescents are better able to address the issue of weight reduction within this treatment modality. Having established the software and treatment process we now wish to perform a randomised, control trial to test the efficacy of this new treatment against that currently provided.

ELIGIBILITY:
Inclusion Criteria:

* Obese children and adolescents aged 10-18

Exclusion Criteria:

Children:

* Having associated learning difficulties
* Who have received medication for associated insulin resistance
* Refusal of parent/legal guardian to give informed consent.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2004-09; Primary Completion 2009-10 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian P Hamilton-Shield, MD, Principal Investigator — University of Bristol and Bristol Royal Hospital for Children
Locations (1):
- Bristol Royal Hospital for Children, Bristol, United Kingdom

REFERENCES:
- [Result] Ford AL, Bergh C, Sodersten P, Sabin MA, Hollinghurst S, Hunt LP, Shield JP. Treatment of childhood obesity by retraining eating behaviour: randomised controlled trial. BMJ. 2009 Jan 5;340:b5388. doi: 10.1136/bmj.b5388. PMID 20051465

RESULTS

PARTICIPANT FLOW:
Groups:
- Allocated to Mandometer Group: Received Mandometer therapy and lifestyle advice.
- Control Arm: Received lifestyle advice alone
Period: Overall Study
Arm/Group | Allocated to Mandometer Group | Control Arm
Started | 54 | 52
Completed | 45 | 46
Not Completed | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Allocated to Mandometer Group (54): Received Mandometer therapy and lifestyle advice.
- Control Arm (52): Received lifestyle advice alone
- Total: Total of all reporting groups
Arm/Group | Allocated to Mandometer Group (54) | Control Arm (52) | Total
Number analyzed (Participants) | 54 | 52 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 54 | 52 | 106
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 12.7 [9.0 to 16.9] | 12.5 [9.1 to 17.5] | 12.6 [9.0 to 17.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 59
  Male | 24 | 23 | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 54 | 52 | 106

OUTCOME MEASURES:

1. Primary Outcome: BMI SDS or Z-score
Description: Body Mass Index standard deviation (s.d.) scores also called Z-scores, are measures of relative weight adjusted for a child's age and sex. In terms of this score for weight management, a lower score would be viewed a beneficial outcome at the end of the intervention. The change in BMI SDS was calculated as the value at 12 months minus value at baseline ( a negative score being beneficial).
Time Frame: 12 months primary/ 18 months secondary outcome
Population: The 12 months data includes Z-score of patients completing study (Mandometer arm n=45, Standard arm n=46) and last recorded Z-score of those withdrawing (Mandometer n=9, Control n=6). At 18 months (6 months after intervention ended) data was available on 44 participants in the active (Mandometer group) and 43 from the control arm.
Measure: Mean (Standard Deviation); unit: Z-Score
Groups:
- Mandometer: Active intervention - one meal eaten per day off Mandometer
  mandometer
  Mandometer: A computerised device, Mandometer, providing real time feedback to participants during meals to slow down speed of eating and reduce total intake; standard lifestyle modification therapy.
Arm/Group | Mandometer | Control
Number analyzed (Participants) | 54 | 52
Z-Score
  Baseline | 3.29 (0.52) | 3.21 (0.45)
  12 months | 2.93 (0.72) | 3.07 (0.56)
  18 months: number analyzed (Participants) | 44 | 43
  18 months | 2.88 (0.74) | 3.07 (0.54)

2. Secondary Outcome: Insulin Sensitivity
Description: Insulin sensitivity was measured by the homeostasis model assessment (HOMA-R) equation: HOMA-R = fasting glucose (mmol/l) × fasting insulin (mIU/l)/22.5. The lower the HOMA-R, the more insulin sensitive the participant is which is considered beneficial to metabolic health.
Time Frame: 12 months
Population: 90 patients completed the intervention study at 12 months. One additional patient withdrew from intervention but agreed to data collection at 12 months. Data unavailable for analysis on one patient allocated to Mandometer.
Measure: Geometric Mean (Full Range); unit: Arbitary units
Arm/Group | Allocated to Mandometer Group (54) | Control Arm (52)
Number analyzed (Participants) | 44 | 46
Arbitary units
  Baseline | 4.04 [0.3 to 15.2] | 4.04 [1.5 to 15.1]
  12 months | 3.27 [0.8 to 13.4] | 3.77 [1.0 to 18.1]

3. Secondary Outcome: Speed Food Consumed
Description: Grams of food eaten per minute in Mandometer® arm compared to standard arm at baseline and 12 months. Reducing speed of eating improves satiety and reduces total food consumed at meals in our overall hypothesis.
Time Frame: 12 months
Population: In only 23 of control cases was baseline data available on eating speed which then could be analysed for change at 12 months.
Measure: Mean (Full Range); unit: gms/min of food consumed
Arm/Group | Allocated to Mandometer Group (54) | Control Arm (52)
Number analyzed (Participants) | 44 | 23
gms/min of food consumed
  Baseline | 29.8 [13.4 to 90.4] | 29.3 [12.6 to 63.9]
  12months | 26.4 [10.2 to 54.8] | 30.6 [12.3 to 54.7]

4. Secondary Outcome: Percentage Body Fat (Measured Using a Tanita Bio-impedance Monitor Model BC-418MA)
Description: Change in % body fat. Calculated as %body fat at end of intervention minus baseline. A negative value being viewed as beneficial outcome.
Time Frame: 12 months
Population: 90 patients completed the intervention study at 12 months. One additional patient withdrew from study but agreed to data collection at 12 months. Data unavailable for analysis on two patients allocated to Mandometer.
Measure: Mean (Standard Deviation); unit: percentage of body fat
Arm/Group | Allocated to Mandometer Group (54) | Control Arm (52)
Number analyzed (Participants) | 43 | 46
percentage of body fat
  Baseline | 43.5 (7.8) | 43 (6.7)
  12 Months | 38.9 (8.5) | 41.6 (6.9)

ADVERSE EVENTS:
Groups:
- Control: Nutritional and activity advice alone
  mandometer
Arm/Group | Mandometer | Control
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/52
Other Adverse Events (participants affected / at risk) | 0/54 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes